CLINICAL TRIAL: NCT03274960
Title: The Effect of Screening and Treatment of Asymptomatic Bacteriuria Every Trimester During Pregnancy on Incidence of Preterm Birth in Harare, Zimbabwe
Brief Title: Screening and Treating Asymptomatic Bacteriuria Every Trimester and Preterm Birth
Acronym: Pretermbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zimbabwe (Other)
Responsible Party: Principal Investigator, Judith Rukweza, DPhil Student, Mrs, University of Zimbabwe
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 127/16/JREC
Record Dates: First submitted 2017-08-25; First posted 2017-09-07 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Preterm Birth; Asymptomatic Bacteriuria in Pregnancy
Keywords: asymptomati bacteriuria, Griess nitrite test, preterm birth
MeSH Terms: conditions — Premature Birth | interventions — Griess reagent; Culture Techniques; Therapeutics

STUDY DESIGN:
Intervention Model Description: The control group shall be receiving the usual current antenatal services which do not include any screening at all for asymptomatic bacteriuria. Control group participants will however be treated as routinely being done when a woman presents with symptoms of a UTI. Control group will therefore continue to get the routine antenatal care service as currently being done at the clinics. Participants in the intervention group will each be screened for asymptomatic bacteriuria once in each trimester using the Griess test. A culture test will be done which will confirm diagnosis of bacteriuria. participants in intervention group who will present with symptoms and who will test positive for bacteriuria with the Griess and culture test will be treated with antibiotics as per usual treatment protocol. A comparison about number of preterm births for intervention group and control group will be done to reveal the effect of the study intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator will not be aware of study group at analysis stage of results. The assessors of outcome will be blinded to study arm as they analyse data to reduce risk of bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Griess, Culture and antibiotic (Experimental): Griess reagents, sulfanilamide and NED added in urine sample for 20 minutes, urine culture using blood agar for 24 hours and treatment with antibiotic every trimester for up to 7 days.
  Interventions: Combination Product: Griess,
- No Griess, culture, treatment (No Intervention): No Griess reagents added in urine sample, no culture test with blood agar and no treatment with antibiotic for every positive results every trimester

INTERVENTIONS:
Combination Product: Griess, — Experimental: Griess, Culture and antibiotic Griess reagents, sulfanilamide and NED added in urine sample for 20 minutes, urine culture using blood agar for 24 hours and treatment with antibiotic every trimester for up to 7 days.
  Other Names: Culture; Treatment
  Arms: Griess, Culture and antibiotic

SUMMARY:
This study is evaluating whether screening of a pregnant woman for asymptomatic bacteriuria in each trimester for early detection and treatment of bacteriuria will reduce the incidence of preterm birth in Harare.

DETAILED DESCRIPTION:
Asymptomatic bacteriuria is common in pregnancy. If the disease is not detected early in pregnancy and treated it often progresses to an acute symptomatic disease, pyelonephritis which is associated with adverse pregnancy outcomes including preterm birth.

It is recommended that every woman be screened for asymptomatic bacteriuria by urine culture test at initial antenatal care visit so that the disease is if identified is treated early to prevent preventable complications of the disease in pregnancy. Culture test is expensive and therefore unavailable at several primary care settings especially in low resource settings where majority of pregnant women register and visit for antenatal care. In Zimbabwe antenatal care at primary care clinics is not including screening for asymptomatic bacteriuria. Majority who present with symptoms are empirically treated.

In this study the Griess nitrite test, an effective inexpensive screening test for asymptomatic bacteriuria is used. the test detects nitrite in urine which is associated with presence of nitrate reducing uropathogens, commonly the gram negative bacteria. All the positive samples will then be further tested by culture for bacteria identification, quantification and antibiotic sensitivity. A Randomized controlled trial research design is being used. participants are randomly allocated to intervention group or control group. Urine samples will be collected and tested 3 times for each recruited participant in the intervention arm. treatment will be initiated for positive result according to sensitivity test. Control group will only be subjected to routine existing antenatal care.

Participants will be recruited before 22 weeks gestation and followed on for second contact by 28 weeks and third contact by 36 weeks. Follow up will be stopped on delivery for noting gestation at delivery, whether preterm or term.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women registering at study site.
* Woman is able to identify her date of last menstrual period.
* Gestation of pregnancy is between 6 and 22 weeks.
* Woman is asymptomatic for bacteriuria
* Woman voluntarily signs the consent form

Exclusion Criteria:

* Pregnant woman ill and unwell
* Pregnant woman unwilling to sign consent form
* Woman who had antibiotic treatment 2 weeks before recruitment
* Woman on long term antibiotic treatment
* Woman who fails to identify date of last menstrual period
* Woman symptomatic for urinary tract infection

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Preterm birth | Preterm birth will be calculated as gestation at birth of baby using date of birth and the first date of last menstrual period.
  Preterm birth will be delivery of a baby before 37 complete weeks of gestation from the first date of last menstrual period. It will be sub-categorized as extremely preterm (<28 weeks), very preterm (28 to <32 weeks) and moderate to late preterm (32 to <37 weeks).

SECONDARY OUTCOMES:
symptomatic bacteriuria | The symptoms will be noted at interviews at follow up after every 6 to 8 weeks from previous contact.
  Noted from history of urinary tract symptoms which include pain on micturition, fever, blood in urine, increased urine frequency, foul smelling urine and cloudy urine.
Isolated uropathogen | These will be available at recruitment by 22 weeks, between 22 and 28 weeks at second screening and at 28 to 36 weeks at the third screening.
  All isolated bacterial species from urine sample identified from culture test. These are bacteria identified to be responsible for asymptomatic bacteriuria.
Antibiotic sensitivity | These will be available at recruitment by 22 weeks, between 22 and 28 weeks at second screening and at 28 to 36 weeks at the third screening
  from urine culture results identified antibiotics sensitive for treatment of isolated bacteria will be noted.
Gestation at birth | Gestation will be calculated at delivery of baby.
  Gestation is the calculated total number of weeks from first date of last menstrual period to the date of delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Muchabaiwa F Gidiri, MD, Study Director — Senior Lecturer, Chairperson Obstetrics and Gynecology Department, University of Zimbabwe; Pasipanodya Nziramasamga, PHD, Study Director — Senior Lecturer, Medical Microbiology Department, University of Zimbabwe; Babil Stray- Pedersen, Professor, Study Director — Doctor, Medisin Department, Oslo University; Clara Haruzivishe, PHD, Study Chair — Senior lecturer, Department of Nursing Science, University of Zimbabwe
Locations (1):
- University of Zimbabwe, Harare, Metropolitan, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
plan to share individual participant information will include sharing culture test results on antibiotic sensitivity for those with positive urine culture results. the in formation shared is intended to assist with effective decision making on selection of the best antibiotic to use to treat asymptomatic bacteriuria.
Supporting Information: Study Protocol, CSR
Time Frame: for the period of study for the protocol As soon as culture results are out
Access Criteria: Soft copy Hard copy